CLINICAL TRIAL: NCT04605315
Title: Indications and Outcomes in Kidney-ureteral Pediatric Lithiasis: Experience of Parma
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Stefania Ferretti, Head of endourology-OU Urology, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 490/2019/OSS*/AOUPR
Record Dates: First submitted 2020-09-30; First posted 2020-10-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Pediatric ALL; Stone, Urinary
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Incidence of paediatric urolithiasis is increasing in Europe and North America. Nowadays the management of stone disease is a common practice in not endemic country. The surgical's treatment is based on similar techniques as for adults. In the last years due to miniaturization of endoscopic instruments endourology has become the best approach to treat urinary stones in children. The investigators have retrospectively reviewed experience from 01/01/2000 to 28/02/2019 in children ≤ 16 years old affected by urinary stones who underwent rigid and flexible ureterorenoscopy and pecutaneous nephrolitotripsy procedures and recorded clinical data, overall success rate and complication.

ELIGIBILITY:
Inclusion Criteria:

* 0-17 yrs old, urinary stones (kidney, ureteral, not bladder), with or without malformations or metabolic diseases

Exclusion Criteria:

* none

Ages: 0 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: 0-17 yrs old, urinary stones (kidney, ureteral, not bladder), with or without malformations or metabolic diseases
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
stone free rate | immediately
  no stones or residual fragment < 4 mm
stone free rate | 3 months follow up
  no stones or residual fragment < 4 mm
complication rate | immediately
  clavien-dindo classification
complication rate | 3 months follow up
  clavien-dindo classification

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Parma, Parma, Italy